CLINICAL TRIAL: NCT07064109
Title: Multi-omics Characterization and Model Construction of Colchicine Anti-inflammatory Therapy Efficacy in Acute Coronary Syndromes Patients
Brief Title: Multi-omics Characterization and Model Construction of Colchicine Anti-inflammatory Therapy Efficacy in ACS Patients
Acronym: MCM-CATE-ACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Xuebo Liu, Director, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJH-2025-07
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: ACS - Acute Coronary Syndrome
Keywords: ACS; colchicine
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine treatment group (Experimental): Adding low-dose colchicine on the basis of standardized treatment
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet Once Daily
- control group (No Intervention): Standardized treatment

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet Once Daily — Colchicine 0.5 MG Oral Tablet Once Daily
  Arms: Colchicine treatment group

SUMMARY:
The aim of this prospective cohort study was to investigate the multi-omics characteristics of the efficacy of colchicine treatment in patients with ACS and to construct a model of efficacy. The main questions the study aims to answer are

- Specific mechanisms of colchicine therapy in patients with ACS; Mechanism-based modelling to identify the population that benefits from colchicine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 80
* ACS (STEMI or NSTE-ACS)
* Patients to receive standardised drug therapy
* Able and willing to provide informed consent

Exclusion Criteria:

* Any contraindication to colchicine or known intolerance to colchicine
* Has been using colchicine for a prolonged period of time for other medical conditions
* Women of childbearing age who are pregnant, breastfeeding or not using effective contraception
* Coronary artery bypass grafting within the last 3 years or planned
* Severe hepatic impairment: elevated serum alanine aminotransferase and/or aminotransferase (ALT) and/or aminotransferase (AST) levels of up to three times the upper limit of normal
* Severe renal impairment: eGFR <30mL/min/1.73m2
* Thrombocytopenia (platelet count less than 100*10⁹/L)
* Active diarrhoea
* Infectious diseases: presence of uncontrollable infectious diseases
* Immune-related diseases: known immune diseases such as systemic lupus erythematosus, asthma, inflammatory bowel disease, gout, malignant tumours, etc.
* Strong CYP3A4 or P glycoprotein inhibitors (e.g., cyclosporine, antiretrovirals, antifungals, erythromycin and clarithromycin) are already in use and no alternative medications can be administered
* Planning to use systemic anti-inflammatory therapies such as NSAIDs, hormones, immunomodulators and chemotherapeutic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of responder | 6 months after enrolment
  1. Resolution of Inflammation: A reduction in high-sensitivity C-reactive protein (hs-CRP) levels to <2.0 mg/L, or a decrease of ≥50% from baseline.
  2. Clinical Stability: No occurrence of major adverse cardiovascular events (MACE), defined as cardiovascular death, non-fatal myocardial infarction, non-fatal ischemic stroke, or urgent revascularization.
  3. Ventricular Remodeling: This is assessed by parameters such as ventricular volume, wall thickness, left ventricular mass, and LVEF (Left Ventricular Ejection Fraction), measured by cardiac magnetic resonance (CMR) or echocardiography.
Number of Participants with Advances in Coronary Artery Physiology and Function | 1 year after enrolment
  Comparing the change in coronary QFR at baseline and one-year follow-up, the sum of QFR of the three major coronary vessels (anterior descending, circumflex, and right coronary artery) was calculated (3V-QFR), and progression in coronary physiology was defined when 3V-QFR minus baseline 3V-QFR at follow-up was ≤ -0.05

SECONDARY OUTCOMES:
Incidence of MACE within one year | 1 year after enrolment
  MACE defined as: death (cardiac or non-cardiac), acute myocardial infarction, stroke, ischaemia-driven haemodialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No